CLINICAL TRIAL: NCT06892678
Title: DFMO Maintenance for Patients With Relapsed/Refractory Ewing Sarcoma or Osteosarcoma
Acronym: DFMO
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-16461
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Osteosarcoma Recurrent; Ewing's Tumor Recurrent
MeSH Terms: interventions — Eflornithine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with DFMO (Experimental): DFMO will be administered orally every 12 hours in 28-day cycles at the FDA approved dosages based on the patient's body surface area (BSA). DFMO tablets are 192 mg.
  * Patients with a BSA < 1.5 m2 will take 768 mg (four tablets) orally twice a day.
  * Patients with a BSA 0.75 to 1.5 m2 will take 576 mg (three tablets) orally twice a day.
  * Patients with a BSA of 0.5 to < 0.75 m2 will take 384 mg (two tablets) orally twice a day.
  * Patients with a BSA of 0.25 to < 0.5 m2 will take 192 mg (one tablet) orally twice a day.
  Interventions: Drug: DFMO

INTERVENTIONS:
Drug: DFMO — DFMO dose will be calculated based on the BSA measured within 14 days prior to the beginning of each cycle. Tablets may be swallowed whole, chewed, or crushed and mixed with soft food or liquid.
  Other Names: Difluoromethylornithine; iWilfin

SUMMARY:
The purpose of this study is to determine the feasibility of administering DFMO to patients with relapsed Ewing sarcoma and osteosarcoma who have completed all planned therapy and have no evidence of disease.

DETAILED DESCRIPTION:
Approximately 30-35% of patients diagnosed with osteosarcoma or Ewing sarcoma will develop relapsed/refractory disease and carry a very poor prognosis. DL-alpha-difluoromethylornithine, commonly known as DFMO or eflornithine, is a synthetic analog of the amino acid ornithine. DFMO has been studied in a number of different cancers as either a therapeutic or a chemopreventative agent and is now FDA approved to reduce the risk of relapse in patients with newly diagnosed high-risk neuroblastoma. As DFMO has now been given to over 100 children with metastatic cancer, dosing and safety in this population is well established. Given the stagnant survival rates for children, adolescents, and young adults with relapsed Ewing sarcoma and osteosarcoma over the past few decades, this study will explore the feasibility of using DFMO in patients with relapsed osteosarcoma and relapsed Ewing sarcoma who are without any evidence of disease at the end of therapy in order to prevent disease recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients < 40 years of age at the time of enrollment
* Diagnosis of relapsed osteosarcoma or relapsed Ewing sarcoma who have completed all planned therapy for their relapse, as described in the protocol, and have no evidence of disease
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1, or 2
* Adequate bone marrow function defined as:
* Peripheral absolute neutrophil count (ANC) greater or equal to 750/microliters
* Platelet count greater or equal to 75,000/microliters (transfusion independent)
* Adequate renal function defined by serum creatinine based on age and gender
* Adequate liver function defined as:
* Total bilirubin ≤ 1.5 x the upper limit of normal (ULN) for age AND
* SGPT (ALT) ≤ 5.0 x ULN for age. For this study the ULN is 45 U/L

Exclusion Criteria:

* Pregnant or breastfeeding females
* Patients must not have an uncontrolled infection
* Patients must not have any significant intercurrent illness

Max Age: 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Administering DFMO | Up to 2 years
  Feasibility will be defined as the ability to successfully administer DFMO to at least 80% of subjects who initiate therapy until either disease recurrence or completion of the maximally allowed duration of therapy. Results will be summarized using basic descriptive statistics.

SECONDARY OUTCOMES:
Event Free Survival | Up to 2 years
  The number/percentage of participants with event-free survival (EFS) will be determined. Event-free survival will be defined as the time from diagnosis until drug discontinuation, disease progression, recurrence at any site, secondary malignancy, death from any cause, or last follow-up, whichever is observed first.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Lee, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Collier AB 3rd, Krailo MD, Dang HM, DuBois SG, Hawkins DS, Bernstein ML, Bomgaars LR, Reed DR, Gorlick RG, Janeway KA. Outcome of patients with relapsed or progressive Ewing sarcoma enrolled on cooperative group phase 2 clinical trials: A report from the Children's Oncology Group. Pediatr Blood Cancer. 2021 Dec;68(12):e29333. doi: 10.1002/pbc.29333. Epub 2021 Sep 8. PMID 34496122
- [Background] Lagmay JP, Krailo MD, Dang H, Kim A, Hawkins DS, Beaty O 3rd, Widemann BC, Zwerdling T, Bomgaars L, Langevin AM, Grier HE, Weigel B, Blaney SM, Gorlick R, Janeway KA. Outcome of Patients With Recurrent Osteosarcoma Enrolled in Seven Phase II Trials Through Children's Cancer Group, Pediatric Oncology Group, and Children's Oncology Group: Learning From the Past to Move Forward. J Clin Oncol. 2016 Sep 1;34(25):3031-8. doi: 10.1200/JCO.2015.65.5381. Epub 2016 Jul 11. PMID 27400942